CLINICAL TRIAL: NCT04655079
Title: Efficacy and Safety of Transcranial dIrect Current stiMulation (tDCS) on Motor and Cognitive Symptoms in Progressive Supranuclear Palsy (PSP) (STIM-PSP)
Brief Title: Efficacy and Safety of Transcranial dIrect Current stiMulation (tDCS) in Progressive Supranuclear Palsy (PSP) (STIM-PSP)
Acronym: STIM-PSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Marina Picillo, Clinical Professor, University of Salerno
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCS 01-2020
Record Dates: First submitted 2020-11-27; First posted 2020-12-04 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Progressive Supranuclear Palsy; Motor and Cognitive Symptoms
Keywords: Progressive Supranuclear Palsy (PSP); Transcranial direct current stimulation (tDCS)
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Neurobehavioral Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be recruited and randomized in two parallel group: group 1 will receive anodal left dlPFC tDCS (real tDCS) and group 2 will receive sham stimulation for 5 days/week for 2 consecutive weeks, in a 2:1 ratio, respectively. Each participant will undergo a clinical evaluation at baseline (T0), immediately after 2 weeks of either real or sham tDCS (T1), at 45-day (T2) and at 3-month follow up (T3) from baseline. PSP phenotypes will be uniformly distributed between treatment arms (ie, =Richardson's syndrome versus non-Richardson's syndrome=1:1).
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization, monitoring and data management will be performed locally. Randomization will be performed using an online list randomizer (random.org). The study coordinator will generate the random allocation sequence before enrollment. Then, one sub-investigator will perform clinical evaluations and another one will administer the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS group (Experimental): Participants receive anodal tDCS on the left dlPFC for 5 days/week for 2 weeks
  Interventions: Device: Anodal transcranial direct current stimulation (a-tDCS)
- Sham group (Sham Comparator): Participants receive sham stimulation on the left dlPFC for 5 days/week for 2 weeks
  Interventions: Device: Sham Condition

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation (a-tDCS) — tDCS is delivered by a battery-driven constant current stimulator thought a pair of saline soaked surface sponge electrodes. The active electrode (anode) is placed on the scalp over the left dlPFC (F3) according to the 10 to 20 international electroencephalogram coordinates) and the cathode is placed over the right deltoid muscle. During real stimulation a constant current of 2mA (milli Ampere) is applied for 20 minutes.
  Other Names: Active tDCS
  Arms: Real tDCS group
Device: Sham Condition — For the sham condition the electrode placement is the same of active tDCS but the electric current is ramped down 5 seconds after the beginning of the stimulation.
  Arms: Sham group

SUMMARY:
This is a double-blind, randomized, sham-controlled clinical trial that aim to verify the safety and the efficacy of anodal transcranial direct current stimulation (tDCS) on cognitive and motor symptoms in Progressive Supranuclear Palsy (PSP) over the left dorsolateral prefrontal cortex (dlPFC).

DETAILED DESCRIPTION:
Progressive Supranuclear Palsy (PSP) is a rapidly progressive neurodegenerative disease characterized by deposition of tau and motor, cognitive and behavioral symptoms. Since no effective treatment is available, non-invasive brain stimulation techniques, such as tDCS, could be a valid complementary therapeutic approach. The tDCS modulates the spontaneous activity of the neural network by applying a direct current flow on the cortical brain areas (anodic or cathodic stimulation). Despite its efficacy in psychiatric disorders, the therapeutic use of tDCS in neurodegenerative diseases requires more systematic studies. The aim of this study is to verify the safety and efficacy of tDCS in PSP on motor, cognitive and behavioral symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PSP according with Movement Disorder Society (MDS) criteria (Hoglinger et al., 2017);
* Age > 40 and < 89 years;
* Presence of a caregiver supportive the patient for all study procedure;
* Ability to walk for at least 5 steps either independently or with a minimum support (another patients holding patient's arm or with a walker)

Exclusion Criteria:

* Presence of electrical stimulators (for example, pacemaker, Deep Brain Stimulation, DBS)
* Difficult in understanding Italian language
* Presence of severe sensory deficits (for example, visual or hearing impairments)
* Education level <5 years
* History of drug abuse
* History of severe psychiatric disorders
* History of transient ischemic attacks
* Cortical or sub-cortical vascular lesions
* Seizures or severe heart problems and previous neurosurgical operations
* Absence of subjective cognitive deficits
* MMSE (Mini-Mental State Examination) score <20
* Left-handedness

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 3-month follow up in verbal fluency task | Baseline (T0); At 3-month (T3)
  fluency in verbal names

SECONDARY OUTCOMES:
Change from baseline to 3-month follow in motor symptoms as assessed with sensor recordings (OPAL system) | Baseline (T0); At 3-month (T3)
  movements recorded with digital sensors (gait and other tasks)
Change from baseline to 3-month follow up in cognitive symptoms as assessed with Montreal Cognitive Assessment (MOCA) | Baseline (T0); At 3-month (T3)
  Cognitive status assessed with Montreal Cognitive Assessment (MOCA). The cut off is 15,5. The minimum value is 0 and the maximum is 30. Higher scores mean a better outcome.
Change from baseline to 3-month follow up in caregiver distress as assessed with Neuropshychiatric Inventory (NPI) | Baseline (T0); At 3-month (T3)
  depression symptoms, apathy, neuropsychiatric symptoms assessed with Neuropshychiatric Inventory (NPI) . The minimum value of distress is 0 and the maximum is 5. Higher scores mean a worse outcome.
Change from baseline to 3-month follow up in executive function as assessed with Frontal Assessment Battery (FAB) | Baseline (T0); At 3-month (T3)
  Executive function assessed with Frontal Assessment Battery (FAB). The cut off is 13,4. The minimum value is 0 and the maximum is 18. Higher scores mean a better outcome.
Change from baseline to 3-month follow up in attention as assessed with Frontal Assessment Battery (FAB) | Baseline (T0); At 3-month (T3)
  Attention assessed with Frontal Assessment Battery (FAB). The cut off is 13,4. The minimum value is 0 and the maximum is 18. Higher scores mean a better outcome.
Change from baseline to 3-month follow up in caregiver distress as assessed with Zarit Carer Burden Burden Interview (ZBI) | Baseline (T0); At 3-month (T3)
  Caregiver distress assessed with Zarit Carer Burden Burden Interview (ZBI). The minimum value is 0 and the maximum is 88. The cut off is 46. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro per le Malattie Neurodegenerative (CEMAND) Dipartimento di Medicina e chirurgia, Sezione Neuroscienze, Università di Salerno, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No